CLINICAL TRIAL: NCT04240054
Title: A Multisite, Phase II Study of Bortezomib, Isatuximab, Cyclophosphamide and Dexamethasone (VICD) Induction in Transplant-Eligible Multiple Myeloma Patients With Renal Insufficiency
Brief Title: Bortezomib, Isatuximab, Cyclophosphamide and Dexamethasone Induction in Transplant-Eligible Multiple Myeloma Patients With Renal Insufficiency
Acronym: VICD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Binod Dhakal, Associate Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00036788
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Renal Insufficiency; Isatuximab
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Bortezomib; isatuximab; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Safety Lead-in Cohort A (Experimental): Six transplant-eligible multiple myeloma patients with renal impairment will be enrolled.
  Bortezomib (1.5 mg/m^2) subcutaneous on days 1,8 and 15 Isatuximab (10 mg/kg) IV on days 1, 8, 15 and 22 Cyclophosphamide (250 mg/m^2) IV on days 1, 8 and 15 Dexamethasone 20 mg PO or IV (10 mg if >75 years) on days 1, 2, 8, 9,15,16, 22 and 23
  Interventions: Drug: Bortezomib; Drug: Isatuximab; Drug: Cyclophosphamide; Drug: Dexamethasone
- Expansion Cohort A (Experimental): 35 transplant-eligible multiple myeloma patients with renal impairment will be enrolled.
  Bortezomib (1.5 mg/m^2)subcutaneous on days 1, 8 and 15 Isatuximab (10 mg/kg) IV on days 1, 8, 15 and 22 Cyclophosphamide (250 mg/m^2) IV on days 1, 8 and 15 Dexamethasone 20 mg PO or IV (10 mg if >75 years) on days 1, 2, 8, 9,15,16, 22 and 23
  Interventions: Drug: Bortezomib; Drug: Isatuximab; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Bortezomib (1.5 mg/m^2) subcutaneous on days 1, 8 and 15
  Other Names: Velcade
Drug: Isatuximab — Isatuximab (10 mg/kg) IV on days 1, 8, 15 and 22
  Other Names: SAR650984
Drug: Cyclophosphamide — Cyclophosphamide (250 mg/m^2) IV on days 1, 8 and 15
  Other Names: Cytoxan; Neosar; cytophosphane
Drug: Dexamethasone — Dexamethasone 20 mg PO or IV (10 mg if >75 years) on days 1, 2, 8, 9, 15, 16, 22 and 23
  Other Names: Baycadron; Decadron; DexPak; TaperDex; Zema-Pak; ZoDex; Zonacort

SUMMARY:
This is a single-arm, open-label phase II study with a safety lead-in phase.

DETAILED DESCRIPTION:
The study hypothesis is that the isatuximab plus bortezomib, cyclophosphamide and dexamethasone (VCD) combination is safe and highly effective even in those with renal insufficiency (RI) from myeloma. In this study, we seek to improve the efficacy of VCD by adding isatuximab in newly diagnosed multiple myeloma patients undergoing autologous stem cell transplant (ASCT) irrespective of renal function.

The primary objective is to determine if the addition of isatuximab to VCD will increase the proportion of subjects achieving very good partial response (VGPR), as defined by the International Myeloma Working Group (IMWG) criteria and by the time of completion of post-ASCT consolidation treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Male or female subjects ≥18 years.
3. Patients must be eligible for high-dose therapy and autologous stem cell transplantation as per institutional guidelines.
4. No prior multiple myeloma (MM) -directed therapy except for dexamethasone (up to 160 mg), bortezomib (up to 5.2 mg/m^2) and/or cyclophosphamide up to 500 mg/m^2 administered for management of acute manifestations of MM (hypercalcemia, renal impairment, pain) for no longer than four weeks prior to enrollment. If subject received any prior therapy, pretreatment parameters necessary for disease characterization and response assessment (at least one of the following: Serum protein electrophoresis (SPEP)/Immunofixation electrophoresis (IFE), 24-hour urine protein with urine protein electrophoresis (UPEP)/ IFE, serum free light chains and bone marrow procedure) must be available.
5. Patients must have documented multiple myeloma as defined by the criteria below (a, b, and c):

   1. Monoclonal plasma cells in the bone marrow of ≥10% or presence of a biopsy proven plasmacytoma AND
   2. Evidence of organ damage or myeloma-defining events (MDE) that can be attributed to the underlying proliferative plasma cell disorder (at least one of the following):

      • Hypercalcemia: corrected serum calcium >1 mg/dL higher than the upper limit of normal (ULN) or >11 mg/Dl.

      OR

      • Anemia: hemoglobin value of >2.0 g/dL below the lower limit of normal, or a hemoglobin value <10.0 g/dL.

      OR
      * Bone marrow plasma cells of >60%. OR
      * Involved/uninvolved light chain ratio ≥100 OR
      * Renal insufficiency: eGFR < 40 mL/min/1.73m^2 (based on the Modification of Diet in Renal Disease MDRD formula). [Cohort A subjects must meet this criterion.] If the patient is enrolled in the renal impaired (RI) A cohort but Cycle 1 Day 1 labs do not meet RI definition, the patient will be considered RI (reconsent and rescreening are not required).
   3. Measurable disease as defined (at least one of the following):

      * Serum M-protein level ≥0.5 g/dL; OR
      * Urine M-protein level ≥200 mg/24 hours; OR
      * Light chain multiple myeloma without measurable disease in the urine: serum immunoglobulin (Ig) free light chains (FLC) ≥10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Female subjects who:

   1. Are postmenopausal for at least one year before the screening visit, OR
   2. Are surgically sterile, OR
   3. Females of childbearing potential or male subjects with female partners of childbearing potential shall be required to use effective contraceptive methods (double barrier method, intrauterine device, oral contraception or abstinence) starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s). A woman is considered of childbearing potential, i.e., fertile, following menarche and until becoming postmenopausal unless permanently sterile. The following highly effective methods of contraception are accepted:

      * Established use of oral, intravaginal, or transdermal combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation.
      * Established use of oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation.
      * Placement of an intrauterine device or intrauterine hormone-releasing system.
      * Barrier methods of contraception: male condom with either cap, diaphragm or sponge with spermicide (double-barrier methods). The use of double-barrier methods should always be supplemented with the use of a spermicide. Female condom and male condom should not be used together.
      * Male sterilization (provided that the partner is the sole sexual partner of the patient and that the sterilized partner has received medical assessment of the surgical success).
      * Sexual abstinence.
      * Female subjects must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
8. Male subjects, even if surgically sterilized (i.e., status postvasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through four months after the last dose of study drug(s) (female and male condoms should not be used together), or
   2. Agree to practice true abstinence during the entire study treatment period from the time of signing the informed consent through 16 weeks after the last dose of study drug(s), when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

1. For renal impaired Cohort A subjects, any subject who requires immediate treatment for management of renal failure (including, but not limited to, dialysis). Such treatment is allowed once the patient becomes stable, based on investigator's discretion.
2. Diagnosed or treated for malignancy other than multiple myeloma, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥3 years before enrollment or documentation that the malignancy required/requires no treatment at time of enrollment.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ (e.g., cervical, breast) with no evidence of disease.
3. Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma.
4. Known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have untreated or active hepatitis C.
5. Concurrent medical condition or disease (e.g., active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study. Specifically, any potential subject who is unsuitable for ASCT would be excluded from the study.
6. Clinically significant cardiac disease, including:

   * Myocardial infarction within six months before Cycle 1, Day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   * Uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] Version 5 Grade 2 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
   * Screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
   * Uncontrolled hypertension.
7. Any of the following laboratory test results at the time of enrollment:

   * Absolute neutrophil count <1.0 × 109/L; no granulocyte colony stimulating factor (G-CSF) treatment in the past seven days are allowed.
   * Hemoglobin level ≤7.5 g/dL (≤5 mmol/L); blood transfusions to maintain hemoglobin >7.5 g/dL are acceptable.
   * Platelet count <75 × 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count <50 × 109/L; no platelet transfusions in the past seven days are allowed.
   * Alanine aminotransferase (ALT) level ≥2.5 × ULN
   * Aspartate aminotransferase (AST) level ≥2.5 × ULN
   * Total bilirubin level ≥1.5 × ULN, (except for Gilbert Syndrome: direct bilirubin ≥2 × ULN)
8. Known allergies, hypersensitivity (if not amenable to premedication with steroids, or H2 blockers), or intolerance to monoclonal antibodies or human proteins, isatuximab or its excipients or known sensitivity to mammalian-derived products.
9. Plasma cell leukemia (>2.0 × 10^9/L circulating plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and/or skin changes), or light-chain amyloidosis.
10. Known or suspected of not being able to comply with the study protocol (e.g., because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
11. Pregnant or breastfeeding or planning to become pregnant starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
12. Plans to father a child starting two weeks before first study drug(s) administration, while on therapy and for 16 weeks following the last dose of study drug(s).
13. Had major surgery within two weeks before Cycle 1, Day 1, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study or within two weeks after the last dose of study drug administration. Note: Subjects with planned surgical procedures to be conducted under local anesthesia are not excluded. Kyphoplasty is not considered a major surgery.
14. Patients with pre-existing uncontrolled pulmonary disease will be excluded; uncontrolled refers to patients having had at least one hospitalization due to pulmonary disease (for example, asthma, chronic obstructive pulmonary disease) within the six months prior to enrollment in the study; patients with previous history of pneumonitis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who achieve very good partial response. | 100 days following autologous stem cell transplant
  This will be measured using the International Myeloma Working Group criteria.

SECONDARY OUTCOMES:
The number of subjects who achieve complete response. | 100 days following autologous stem cell transplant.
  This will be measured using the International Myeloma Working Group criteria.
The number of subjects who achieve partial response. | 100 days following autologous stem cell transplant.
  This will be measured using the International Myeloma Working Group criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No